CLINICAL TRIAL: NCT07152444
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Ascending Doses of QLS1410 in Healthy Chinese Adults and Participants With Mild Essential Hypertension
Brief Title: A Phase I Trial of QLS1410 in Healthy Chinese Adults and Participants With Mild Essential Hypertension
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QSL1410-101
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS1410 (Experimental): Part A: Healthy adults will be randomized (6:2) to receive a single dose (1.5 mg ~ 20 mg) of QLS1410 or placebo,especially, the starting dose will be 0.5 mg of QLs1410
  Part B: QLS1410 will be administered under the fasted or fed conditions in two different periods separated by a wash-out interval of 14 days. The dose of QLS1410 or placebo is based on upcoming data from SAD part.
  Part C: Hypertensive participants will be randomized (8:2) to receive QLS1410 or placebo QD for 14 continuous days. The starting dose of QLS1410 or placebo is based on upcoming data from SAD part.
  Interventions: Drug: QLS1410 (CYP11B2 inhibitor)
- Placebo (Placebo Comparator): Part A: Healthy adults will be randomized (6:2) to receive a single dose (1.5 mg ~ 20 mg) of QLS1410 or placebo
  Part B: QLS1410 will be administered under the fasted or fed conditions in two different periods separated by a wash-out interval of 14 days. The dose of QLS1410 or placebo is based on upcoming data from SAD part.
  Part C: Hypertensive participants will be randomized (8:2) to receive QLS1410 or placebo QD for 14 continuous days. The starting dose of QLS1410 or placebo is based on upcoming data from SAD part.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: QLS1410 (CYP11B2 inhibitor) — QLS1410 tablets
  Arms: QLS1410
Drug: placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and food effect of single and multiple ascending doses of QLS1410 in healthy Chinese adults and participants with mild essential hypertension

DETAILED DESCRIPTION:
This study consists of three parts, as follows:

Part A is a randomized, placebo-controlled, double-blind single ascending dose (SAD) study in healthy Chinese adults, consisting of 5 cohorts. Starting dose of 0.5 mg by oral administration are planned. Once sufficient safety and PK data are obtained from the SAD cohorts, the SMC will determine the dosage of initial cohort in Part B and Part C.

Part B is a randomized, open-label, two-cycle, crossover food effect (FE) study under fasting and fed (high-fat meal) conditions.

Part C is a randomized, placebo-controlled, double-blind multiple ascending doses (MAD) study in participants with mild essential hypertension, consisting of 3 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Part A & Part B: Healthy Participants
* Able to understand and willing to comply with all study visits, procedures, restrictions and provide the written informed consent form (ICF).
* Males and females aged 18 to 55 years, inclusive.
* Weight ≥ 50 kg for males and ≥ 45 kg for females, Body mass index (BMI) between 18 and 26 kg/m^2, inclusive, at screening.
* Has a mean seated office systolic blood pressure (SBP) 110~139 mmHg (inclusive) and diastolic blood pressure (DBP) 70~89 mmHg (inclusive) at screening and baseline; measured 3 times consecutively (1-2 min intervals).
* QTcF (QT corrected using Fridericia's formula) <450 ms for males and <470 ms for females.
* Participants (including partners) must agree to abstain from sperm/egg donation and pregnancy plans, and to use highly effective contraception, from signing the ICF until 3 months after receiving the last dose of investigational product.
* Part C: Participants with Mild Essential Hypertension
* Able to understand and willing to comply with all study visits, procedures, restrictions and provide the ICF.
* Males and females aged 18 to 65 years (18 to 65 years in MAD study), inclusive.
* Weight ≥ 50 kg for males and ≥ 45 kg for females, BMI between 18 and 28 kg/m^2, inclusive, at screening.
* Has a mean seated office SBP 140~159 mmHg (inclusive) and DBP 85~99 mmHg (inclusive) at screening and baseline; measured 3 times consecutively (1-2 min intervals).
* QTcF <450 ms for males and <470 ms for females.
* No use of antihypertensive medications (including ACEIs, ARBs, CCBs, ARNIs, diuretics, etc.) within 30 days prior to signing the ICF.
* Participants (including partners) must agree to abstain from sperm/egg donation and pregnancy plans, and to use highly effective contraception, from signing the ICF until 3 months after receiving the last dose of investigational product.

Exclusion Criteria:

* Part A & Part B: Healthy Participants
* Any medical condition/disease at screening deemed by the investigator to require exclusion, including but not limited to the nervous, psychiatric, cardiovascular, hematologic/lymphatic, immune, respiratory, digestive, urinary, metabolic and skeletal systems.
* Dysphagia or any surgical condition/disease that may affect drug absorption, distribution, metabolism, or excretion, at screening.
* Use of systemic corticosteroids within 3 months prior to screening.
* Mean pulse/heart rate (HR) >100 or <50 bpm after ≥5 min of rest at screening (measured 3 times consecutively).
* Any laboratory abnormalities that meet the test requirements should be noted during screening (if necessary, retest can be conducted at least one week apart):
* Smoking >5 cigarettes/day on average within 6 months before screening, or current use of e-cigarettes.
* Alcohol consumption >14 units/week (1 unit = 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine) within 6 months before screening, or has a positive breath alcohol test at screening.
* Blood donation >400 mL within 3 months or >200 mL within 4 weeks before screening, or plan to donate blood during the study.
* Use of strong CYP3A4 or CYP1A2 inhibitors within 7 days or 5 half-lives (whichever is longer) before screening. Use of strong CYP3A4 inducer within 14 days or 5 half-lives (whichever is longer) before screening.
* Use of any prescription drugs, OTC drugs, traditional medicines, and dietary supplements within 2 weeks or 5 half-lives (whichever is longer) prior to randomization.
* Pregnant/lactating females or positive pregnancy test at screening.
* Inability to tolerate a high-fat meal (for Part B only).

Part C: Participants with Mild Essential Hypertension

* Secondary hypertension.
* Orthostatic tachycardia or hypotension at screening, or history of related symptoms (e.g., dizziness, weakness, blurred vision upon standing).
* History of syncope.
* Metabolic/cardiovascular disorders: 1) Diabetes (fasting glucose ≥7.0 mmol/L [126 mg/dL] or HbA1c ≥6.5%); 2) History of cardiovascular events (e.g., stroke, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention, heart failure hospitalization) or clinically significant valvular disease; 3) Personal/family history of long QT syndrome, torsades de pointes (TdP), arrhythmias, or sudden cardiac death; 4) Other conditions that may interfere with the study or increase risk, per investigator judgment.
* Laboratory abnormalities (as defined in Part A/B, with repeat testing allowed).
* Any other condition deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events as assessed by CTCAE v5.0 | up to approximately 1 month

SECONDARY OUTCOMES:
Area under the curve plasma concentration from time zero to last measurable concentration [AUC(0-last)] | up to approximately 1 month
Area under the curve plasma concentration from time zero to infinity [AUC(0-∞)] | up to approximately 1 month
Maximum observed plasma concentration (Cmax) | up to approximately 1 month
Terminal elimination half-life (t1/2) | up to approximately 1 month
Apparent clearance (CL/F) | up to approximately 1 month
Apparent volume of distribution (Vz/F) | up to approximately 1 month
Mean residence time (MRT) | up to approximately 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China